CLINICAL TRIAL: NCT05660122
Title: A Multi-Center, Prospective, Observational Study to Evaluate the Improvement Effect on Subjective Symptom of FEXUCLUE Tab. in Patients With Erosive Gastroesophageal Reflux Disease
Brief Title: A Study to Evaluate the Improvement Effect on Subjective Symptom of FEXUCLUE Tab
Status: Completed | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWFE_P405
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: patients with gastroesophageal reflux disease
  Interventions: Drug: Fexuprazan Hydrochloride

INTERVENTIONS:
Drug: Fexuprazan Hydrochloride — Fexuclue Tablet 40mg
  Other Names: Fexuclue Tablet

SUMMARY:
This observation study is a large-scale, prospective, and multi-organ observation study to observe the improvement effect of the self-evaluation results (PRO) of erosive gastroesophageal reflux disease at least 4 to 8 weeks after administration of Fexuclue Tab.

DETAILED DESCRIPTION:
This observation study is a large-scale, prospective, and multi-organ observation study to observe the improvement effect of the self-evaluation results (PRO) of erosive gastroesophageal reflux disease at least 4 to 8 weeks after administration of Fexuclue Tab.

Subjects who met the inclusion/exclusion criteria will administer Fexuclue Tablet once a day for four weeks after registration, regardless of their meals. If esophagitis is not treated or symptoms continue after 4 weeks of administration, the subject will continue to administer Fexuclue Tablet for 4 more weeks (maximum administration period: 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged 19 to 75 years of age at the time of registration.
2. A patient with erosive gastroesophageal reflux disease who is scheduled to administer Fexuclue Tab. for the first time based on the medical judgement of the researcher based on the medication authorization.
3. A person who voluntarily agrees to participate in this observation study and signed the informed consent form.

Exclusion Criteria:

1. A person who falls under the prohibition of administration according to the permission for Fexuclue Tablet

   * Patients with hypersensitivity to the components of Fexuclue tablet or Fexuclue tablet and a history thereof
   * Patients undergoing Atazanavir, Nelfinavir or Lilpivirin-containing preparations
   * Pregnant and lactating women
   * Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabortion
2. A person who participates in another clinical trial and is administering (applying) clinical trial drugs or clinical trial medical devices;
3. In addition to the above, a person who has determined that the researcher (the doctor in charge) is not suitable for participation in this observation study

Ages: 19 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This observation research plan assumes the following.
  1. level of signification, α=0.05
  2. Distance from Mean to Limits = 0.067
  3. Standard deviation of the amount of change at the time of two weeks compared to the baseline of the RDQ score = 1.66
  As a result of calculating using PASS2020 based on the above assumptions, the number of study subjects required to conduct this study was 2,359. In consideration of the dropout rate of about 20% in the calculated results, we intend to recruit 3,000 study subjects.
Sampling Method: Non-Probability Sample
Enrollment: 2852 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Average score change in RDQ | at 4 weeks (up to 8 weeks)
  Average score change in RDQ at 4 weeks (up to 8 weeks) from baseline

SECONDARY OUTCOMES:
Average individual score change in RDQ | at 4 weeks (up to 8 weeks)
  Average individual score change in RDQ at 4 weeks (up to 8 weeks) from baseline
RDQ validity rate | at 4 weeks (up to 8 weeks)
  RDQ validity rate at 4 weeks (up to 8 weeks) from baseline
Overall improvement evaluated by the subjects | at 4 weeks (up to 8 weeks)
  Overall improvement evaluated by the subjects at 4 weeks (up to 8 weeks) from baseline
Overall improvement evaluated by the researchers | at 4 weeks (up to 8 weeks)
  Overall improvement evaluated by the researchers at 4 weeks (up to 8 weeks) from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Undecided